CLINICAL TRIAL: NCT00010777
Title: Fibromyalgia: A Randomized Controlled Trial of a Mind/Body Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: P50AT000084-01P2 (NIH); P50AT000084-01 (NIH); NCT00009152 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

INTERVENTIONS:
Procedure: Multiple Component Mind/Body therapy

SUMMARY:
The goal of this proposal is to evaluate the efficacy of a multiple component mind-body (MCMB) therapy for fibromyalgia, both in short and long term outcomes. Preliminary work suggests that FM patients do benefit from MCMB therapy (Singh et al 1998; Creamer et al 1998). This two-arm clinical trial will randomize 110 patients to either a 12 week MCMB intervention or a 12 week education/attention intervention. The primary aims of this study are 1) to determine if a 12 week MCMB intervention improves short term (i.e. at 12 weeks) outcomes in FM patients compared to an education/attention control group; and 2) to determine if a 12 week MCMB intervention improves long term (i.e. at 24 weeks) outcomes in FM patients compared to an education/attention control group.

A secondary aim of this project involves determining if there are patient characteristics (i.e. disease severity and duration, demographics, psychological factors) associated with improvements in short or long term outcomes as well as responses to the MCMB intervention.

The primary outcome measure will include physical functioning and pain as measured by the Fibromyalgia Impact Questionnaire.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a common, complex and chronic condition of unknown etiology (Carette 1994). It is characterized by widespread musculoskeletal pain, multiple tender points, fatigue and a range of other symptoms (Wolfe 1990). FM accounts for 15% of rheumatology consultations, with a prevalence of 2% in the general population (3.4% in females and 0.5% in males), rising to 7% in the elderly females (Wolfe 1995). Disability levels in social and work roles, as well as use of medical care, is high. Current treatment options often meet with limited success.

The goal of this proposal is to evaluate the efficacy of a multiple component mind-body (MCMB)therapy for fibromyalgia, both in short and long term outcomes. Preliminary work suggests that FM patients do benefit from MCMB therapy (Singh et al 1998; Creamer et al 1998). This two-arm clinical trial will randomize 110 patients to either a 12 week MCMB intervention or a 12 week education/attention intervention. The primary aims of this study are (1) to determine if a 12 week MCMB intervention improves short term (i.e. at 12 weeks) outcomes in FM patients compared to an education/attention control group; and (2) to determine if a 12 week MCMB intervention improves long term (i.e. at 24 weeks) outcomes in FM patients compared to an education/attention control group.

A secondary aim of this project involves determining if there are patient characteristics (i.e. disease severity and duration, demographics, psychological factors) associated with improvements in short or long term outcomes as well as responses to the MCMB intervention.

The primary outcome measure will include physical functioning and pain as measured by the Fibromyalgia Impact Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fibromyalgia by patient's own health care provider
* ACT classification of fibromyalgia verified by rheumatological examination: a) widespread pain (axial plus upper and lower segment plus left-and-right-sided pain for 3 months or longer; b) tenderness at 11 or more of the 18 specific tender point sites
* Read and speak English fluently
* Be able to attend group intervention session if assigned to that group
* Able to give informed consent

Exclusion Criteria:

* Pregnancy
* Substance abuse
* Major psychiatric disorder (that would prevent compliance)
* Involvement in impending litigation or judgment for disability workmen's compensation
* Uncontrolled hypertension, uncontrolled diabetes, congestive heart failure or other severe chronic medical conditions judged by the clinician to place the patient at risk of possible severe consequences of their disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Brian Berman, Principal Investigator — Univ. of Maryland/Complementary Medicine Program

REFERENCES:
- [Background] Astin JA, Berman BM, Bausell B, Lee WL, Hochberg M, Forys KL. The efficacy of mindfulness meditation plus Qigong movement therapy in the treatment of fibromyalgia: a randomized controlled trial. J Rheumatol. 2003 Oct;30(10):2257-62. PMID 14528526